CLINICAL TRIAL: NCT02091492
Title: Teriparatide for Fracture Repair in Humans: A Prospective, Randomized, Double-blind Placebo-controlled Pilot Study in Female and Male Patients With Proximal Humerus Fracture: The TERAFRAP Study
Brief Title: Teriparatide for Fracture Repair in Humans
Acronym: TERAFRAP
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: no participants
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Christian Muschitz, Senior Consultant for Internal Medicine, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Vinforce_006; # 317.276.2000 (Other Grant/Funding Number: Eli Lilly and Company, Lilly Corporate Center, Indianapolis, IN 46285, USA)
Record Dates: First submitted 2014-03-13; First posted 2014-03-19 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-09

CONDITIONS: Osteoporosis, Age-Related; Humeral Fractures
Keywords: Proximal humerus fracture, teriparatide
MeSH Terms: conditions — Osteoporosis; Humeral Fractures | interventions — Teriparatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Teriparatide (Active Comparator): Teriparatide 20µg daily subcutaneous injection for 12 weeks after proximal humerus fracture
  Interventions: Drug: Teriparatide
- Placebo-Teriparatide (Placebo Comparator): Placebo-Teriparatide 20 µg daily subcutaneous injection for 12 weeks after proximal humerus fracture
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Teriparatide — Teriparatide 20 µg sc (subcutaneous injection) each day for 12 weeks
  Other Names: Forteo
  Arms: Teriparatide
Drug: Placebo — Placebo teriparatide sc (subcutaneous injection) each day for 12 weeks
  Arms: Placebo-Teriparatide

SUMMARY:
This study will test the hypothesis that daily subcuaneous administration of 20µg of teriparatide (TPTD) as compared to daily subcuaneous placebo for twelve weeks accelerates proximal 2-segment humerus fracture healing and improves the three dimensional structural properties of bone as measured via quantitative bone image analysis and finite element modeling assessed by quantitative computed tomography.

DETAILED DESCRIPTION:
1. Primary objective:

   The primary objective is the quantitative assessment of fracture healing (2-segment proximal humerus frafcture) in the treatment (daily teriapratide 20µg subcitaneous injection for 12 weeks) and in the placebo group (daily placebo subcutaneous injection for 12 weeks) based on computed tomography data (QCT; baseline and after 12 weeks) and computational analysis of the three simensional bone structure in the fracture zone. Bone structure will be assessed by means of quantized bone texture characteristics (callus formation, improvement of trabecualar and cortical bone structure) in the vicinity of the fracture.
2. Secondary objectives:

2.1.Detection and quantification of changes in bone mineralization at the fracture site between a baseline QCT scan and a follow-up QCT scan (planned interval: 12 weeks) using 3-D texture-based cluster analysis between the two groups.

2.2 Evaluation of bone strength variation in the proximal humerus and the measurement of biomechanical properties (stiffness, strength, damage) based on the Finite Element (FE) technique between the two groups.

2.3.Baseline characterization of osteoporotic study population: age, sex, concomitant diseases, serum markers of bone formation and bone resorption, serum colecalciferol levels.

2.4.Evaluation of fasting bone formation and resorption markers at baseline and after 3 months follow up between the TPDT and the placebo group.

2.5.Assessment of quality of life improvement for TPTD and placebo groups with EQ-5D questionnaire (measurement every 4 weeks).

2.6.Assessment of pain reduction in TPTD and placebo groups by visual analog scale (VAS) during 12 weeks (measurement every 4 weeks).

2.7.Assessment of functional testing after 3 and 6 months (functional testing score (ASES Score: "American Shoulder and Elbow Surgeon Score")

2.8.Dual energy x-ray absorptiometry (DXA) bone mineral density (BMD) measurements of lumbar spine and early changes of geometrical hip parameters (cross sectional area - CSA, cross sectional moment of inertia - CSMI), hip BMD(femoral neck and total hip area) and total body (lean mass, fat mass, total body BMD)

2.9. Number of Participants with Adverse Events as a Measure of Safety and Tolerability

ELIGIBILITY:
Inclusion Criteria:

* recent proximal 2-segment humerus fracture (0-8 days post fracture)
* no surgical treatment at fractured site
* signed informed consent
* postmenopausal female and male patients aged 60 - 85 years
* established osteoporosis as defined by BMD measured with DXA-technology (dual energy X-ray absorptiometry) with a T-score ≤ -2.0 spine or hip

Exclusion Criteria:

* Hypersensitivity to the active substance or to any of the excipients.
* Pre-existing hypercalcemia
* Severe renal impairment (eGFR< 35ml/min)
* Metabolic bone diseases (including hyperparathyroidism and Paget's disease of the bone) other than primary osteoporosis or glucorticoid-induced osteoporosis.
* Unexplained elevations of alkaline phosphatase
* Prior external beam or implant radiation therapy to the skeleton
* Patients with skeletal malignancies or bone metastases should be excluded from treatment with teriparatide.
* any prior antiresorptive therapy (oral/intravenous bisphosphonates, RANKL-antibody, SERMs)
* any prior strontium ranelate therapy
* any prior TPTD of PTH 1-84 therapy
* malignancies ≤ 5 years except basalioma
* hypo-/hypercalcemia
* baseline 25-OH vitamin D3 level ≤10 ng/ml
* prosthesis at fractured and contralateral humerus

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-06; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Identification of bone and callus patterns in the CT data at the fracture site | 12 weeks
  As a basis for change quantification, we will identify 3D micro-architecture patterns that occur in the study CT data. These patterns are either learned based on annotated examples, manual segmentation of specific regions in a number of reference examples, or in a data-driven fashion (computer based identification of pattern classes).

SECONDARY OUTCOMES:
Finite Element Analysis (FEA) of QCT (quantitative computed tomography) data | 12 weeks
  The FEA Method will be a second diagnostic tool in order to evaluate the change in bone strength in the proximal humerus during treatment.

OTHER OUTCOMES:
Tracking geometry during bone healing | 12 weeks
  The extent of bridging and callus formation will be quantified, based on the voxel-wise comparison of follow-up data. The accumulated density difference between baseline and follow-up over a region of interest serves as parameter.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Muschitz, M.D., Principal Investigator — Medical University Vienna, St. Vincent Hospital Vienna, Austria
Locations (1):
- Medical University Vienna; St. Vincent Hospital, Vienna, Vienna, Austria

REFERENCES:
- [Background] Aspenberg P, Johansson T. Teriparatide improves early callus formation in distal radial fractures. Acta Orthop. 2010 Apr;81(2):234-6. doi: 10.3109/17453671003761946. PMID 20367417